CLINICAL TRIAL: NCT00477685
Title: Study of the Safety and Effectiveness of the OculusGenTM Collagen Matrix Implant as an Aid in Phacotrabeculectomy Surgery
Brief Title: Ologen (OculusGen)-Phacotrabeculectomy Historical Control Study in India
Status: Completed | Type: Observational
Sponsor: Pro Top & Mediking Company Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: Mediking 0704; OculusGen-2007-04-20 (Other: Aeon Astron Europe B.V.)
Record Dates: First submitted 2007-05-23; First posted 2007-05-24 (Estimated); Results first posted 2012-03-29 (Estimated); Last update posted 2017-08-14 (Actual); Status verified 2017-07

CONDITIONS: Glaucoma; Cataract
Keywords: Glaucoma; Collagen matrix; OculusGen; Phacotrabeculectomy; anti scarring; tissue engineering; ologen; Aeon Astron
MeSH Terms: conditions — Glaucoma; Cataract

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months

GROUPS / COHORTS (1):
- OculusGen Collagen Matrix: OculusGen Biodegradable Collagen Matrix Implant in Trabeculectomy.
  Interventions: Device: OculusGen Biodegradable Collagen Matrix Implant

INTERVENTIONS:
Device: OculusGen Biodegradable Collagen Matrix Implant — OculusGen Biodegradable Collagen Matrix Implant in Trabeculectomy.

SUMMARY:
1. . Study Objective: The objective of this study is to determine the safety and effectiveness of the OculusGenTM Biodegradable Collagen Matrix Implant in phacotrabeculectomy surgery. The primary endpoint is to prove the effectiveness via the reduction of Intraocular Pressure, and the secondary endpoint is to prove the safety via the incidence of complications and adverse events.
2. . Study Design: The study is designed as a historical controlled study. Patient who meet the inclusion/exclusion criteria and sign the informed consent form will be included for this study. The allocation of subjects is non-randomized, and there is a single group for assignment.
3. . Follow-Up: This investigation is including 7 post-operative visits and follow-up within 6 months from the date of surgery. Patients should be seen at postoperative days 1, 7, 14, 30, 60, 90 and 180. The visit window of ± 7 days is allowed for the 30, 60, 90 and 180 day visits. The further follow-up of subject after trial is continually tracked by the investigator.

DETAILED DESCRIPTION:
ologen collagen matrix is applied for the phacotrabec surgery.

ELIGIBILITY:
Subject inclusion criteria:

1. Age 18 years or over.
2. At least one eye diagnosed with glaucoma and receiving maximally tolerated medical therapy.
3. Visually significant cataract with visual acuity of less than or equal to 6/12.
4. Subject able and willing to cooperate with investigation plan.
5. Subject willing to sign informed consent form.

Subject exclusion criteria:

1. Known allergic reaction to collagen.
2. Subject is on Warfarin and discontinuation is not recommended.
3. Subject with normal tension glaucoma or aphakic glaucoma.
4. Subject with corneal disease.
5. Participation in an investigational study during the 30 days proceeding phacotrabeculectomy.
6. Ocular infection within 14 days prior to phacotrabeculectomy.
7. Pregnant or breast-feeding women.
8. Monocular subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 10
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2007-05; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: SPS Grewal, MD, Principal Investigator — Grewal Eye Institute
Locations (1):
- Grewal Eye Institute, Chandigarh, India

REFERENCES:
- [Result] Chen HS, Ritch R, Krupin T, Hsu WC. Control of filtering bleb structure through tissue bioengineering: An animal model. Invest Ophthalmol Vis Sci. 2006 Dec;47(12):5310-4. doi: 10.1167/iovs.06-0378. PMID 17122118
- [Result] Hsu WC, Spilker MH, Yannas IV, Rubin PA. Inhibition of conjunctival scarring and contraction by a porous collagen-glycosaminoglycan implant. Invest Ophthalmol Vis Sci. 2000 Aug;41(9):2404-11. PMID 10937547

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | OculusGen Collagen Matrix
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | OculusGen Collagen Matrix
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 3
Region of Enrollment [Number; unit: participants]
  India | 10

OUTCOME MEASURES:

1. Secondary Outcome: Number of Participants With Any Complications or Adverse Events.
Description: Observation of the incidence of complications, including transient shallow anterior chamber, hyphema, choroidal detachment, hypotony or endophthalmitis.
Time Frame: 180 day
Measure: Number; unit: participants
Arm/Group | OculusGen Collagen Matrix
Number analyzed (Participants) | 10
participants | 0

2. Primary Outcome: Preoperative and Postoperative Intraocular Pressure
Description: The preoperative and postoperative intraocular pressure is measured as mmHg at baseline and 90 days.
Time Frame: baseline and 90 days
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | OculusGen Collagen Matrix
Number analyzed (Participants) | 10
mm Hg
  Preoperative intraocular pressure | 20.1 (8.02)
  Postoperative intraocular pressure | 9 (3.32)
Statistical Analysis 1: Comparison: OculusGen Collagen Matrix; Null hypothesis: the postoperative intraocular pressure at 90 days equals the preoperative intraocular pressure at baseline; Test type: Superiority or Other; p = 0.01, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Up to 90 days after surgery.
Description: To assess if there was any complications or adverse events, including shallow anterior chamber, hyphema, choroidal detachment, hypotony or endophthalmitis in any patients.
Arm/Group | OculusGen Collagen Matrix
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

LIMITATIONS AND CAVEATS:
Limited sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No